CLINICAL TRIAL: NCT05027867
Title: An Open-Label, Multicenter, Phase 2 Study of the Safety and Efficacy of KRT-232 in Subjects With Relapsed or Refractory Small Cell Lung Cancer (SCLC)
Brief Title: KRT-232 in Subjects With Relapsed or Refractory Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unanticipated and extremely high screen failure rate. There was no evidence of safety concerns in the study.
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-112
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma; Small Cell Lung Cancer Extensive Stage; Small Cell Lung Cancer Recurrent
Keywords: navtemadlin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): KRT-232 240 mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232
- Arm 2 (Experimental): KRT-232 180 mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232

INTERVENTIONS:
Drug: KRT-232 — Administered by mouth
  Other Names: navtemadlin

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, for the treatment of patients with relapsed or refractory small cell lung cancer.

This study will be conducted in 2 parts. Part 1 will evaluate two treatment arms, each with a different KRT-232 dose. Part 2 will continue the evaluation of the selected treatment arms from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of SCLC documented as TP53WT
* Disease must be measurable per RECIST Version 1.1
* Evidence of radiographic progression during or after at least one prior platinum-containing therapy with no curative therapy available. Subjects who have received only one prior line of therapy must not be candidates for platinum-based regimens at relapse.
* Subjects must have received a checkpoint inhibitor (PD-1 or PD-L1) unless contraindicated if checkpoint inhibitors are approved and available.
* ECOG ≤ 2

Exclusion Criteria:

* Symptomatic or uncontrolled central nervous system (CNS) metastases.
* Prior treatment with MDM2 inhibitors
* Chemotherapy, immune therapy, cytokine therapy, or any investigational therapy within 14 days prior to the first dose of study treatment
* Grade 2 or higher QTc prolongation (> 480 milliseconds per NCI-CTCAE criteria, version 5.0)
* History of major organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) of each arm | 24 weeks
  The proportion of subjects achieving partial response or better per RECIST 1.1

SECONDARY OUTCOMES:
Duration of response (DOR) of each arm | 1 year
  Time from initiation of response to disease progression or death
Progression-free survival (PFS) of each arm | 1 year
  Time from first dose to disease progression or death
Overall survival (OS) of each arm | 1 year
  Time from first dose to death
Disease control rate (DCR) of each arm | 24 weeks
  The proportion of subjects achieving stable disease or better per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (33):
- United States (9):
  - Florida Cancer Specialists - 3840 Broadway, Fort Myers, Florida
  - Florida Cancer Specialists - 560 Jackson St, Suite 220, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mark H Zangmeister Center - 3100 Plaza Properties Boulevard, Columbus, Ohio
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
- Flinders Medical Centre, Bedford Park, South Australia, Australia
- France (8):
  - Centre Hospitalier de Mulhouse - Hopital Emile Muller, Mulhouse, France/Haut-Rhin
  - Edog - Ico - Ppds, Angers, Maine-et-Loire
  - Hôpital Louis Pradel, Bron, Rhône
  - Hospices Civils de Lyon, Lyon, Rhône
  - Hôpital de La Croix Rousse, Pierre-Bénite, Rhône
  - EDOG - Institut Bergonie - PPDS, Bordeaux
  - CHU de Grenoble, Grenoble
  - Hopital Nord AP-HM, Marseille
- Germany (3):
  - Klinik für Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar, Baden-Wurttemberg
  - Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Evangelische Lungenklinik Berlin, Berlin
- Bacs Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county, Hungary
- South Korea (2):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
- Spain (9):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitario 12 de Octubre, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Clinica Universidad Navarra - Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia